CLINICAL TRIAL: NCT00469924
Title: Effect of an Automated Paging System on Response to Critical Laboratory Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Edward Etchells, Associate Professor, Staff Physician, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Etchells1
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Critical Laboratory Values; Drug Laboratory Interactions; Drug Drug Interactions
Keywords: Informatics; Clinical Laboratory Information Systems; Hospital Communication Systems; Laboratory Techniques and Procedures; Point-of-Care Systems; Therapy, Computer-Assisted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alerting system ON (Experimental): Alerting system is ON
  Interventions: Procedure: Real Time Clinical Alerting
- Alerting system OFF (No Intervention): Alerting system is OFF

INTERVENTIONS:
Procedure: Real Time Clinical Alerting
  Arms: Alerting system ON

SUMMARY:
Patients in hospitals may develop serious problems that are detected by blood tests. It is very important for the physicians to be notified of these abnormal blood tests as soon as possible. Currently, this is done using phone calls from the lab to the nurse. The nurse then pages the doctor and waits for a call back. We are conducting a study using an automated paging system that immediately alerts the physician directly. We will test whether the automated system affects the time for the physician to respond to the abnormality. If the physician's patient has a serious laboratory result, we will automatically send this laboratory result to the physician's PDA. We will also provide guidelines for treating the patient. These guidelines will come from existing hospital policies where available, or from local expert opinion. We will determine whether patients get better and faster care because of the automated alerting system.

DETAILED DESCRIPTION:
We will evaluate the effect of real time clinical alerting on the time to response and the quality of the response to critical laboratory values. We define time to response as the time from acceptance of the laboratory value in the laboratory information system to the time that a physician's order is written in response to the laboratory value. In the absence of a timed physician order, we use the time of administration of treatment to estimate the time of response. We define the quality of response as whether the treatment was consistent with existing hospital policies and expert guidelines.

This will be a prospective interrupted time series study.

The setting is secondary-tertiary care inpatient general medicine units at academic teaching hospitals (Sunnybrook and UHN). The physician participants are staff physicians and medical residents in the Division of General Internal Medicine. The patient participants are general internal medicine inpatients with critical laboratory values. The intervention is an automated real time clinical alerting system that includes evidence based decision support and patient specific information about critical laboratory abnormalities. There are two primary outcome measures: (1) time to response, defined as the time from the critical laboratory abnormality to time of resolution of the critical laboratory abnormality, and (2) quality of response, defined as whether the response was concordant with existing evidence based protocols of care. Secondary outcome measures will be: length of stay, mortality, time to resolution of the abnormality, and frequency of recurrence of the abnormality. Other process measures will be: quality of response, time to resolution, and proportion resolved within 24 hours. Time to response is defined as time from the identification of the critical value in the laboratory to time of a physician order in response to the abnormality.

There are two primary outcome measures: (1) time to response, defined as the time from the critical laboratory abnormality to time of a physian order in response to the critical laboratory abnormality, and (2) quality of response, defined as whether the response was concordant with existing evidence based protocols of care. Secondary outcome measures will be: length of stay, mortality, time to resolution and frequency of recurrence. Time to resolution is the time from the initial laboratory abnormality to the time that the abnormality resolves. Frequency of recurrence is the proportion of patients who develop a second episode of the same critical abnormality after resolution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with critical laboratory values or hazardous drug-lab or drug-drug conditions, admitted to inpatient general medicine units

Exclusion Criteria:

* Values or conditions where no clinical action can be taken

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
(1) time to response, defined as the time to a physician order and (2) quality of response, defined as whether the response was concordant with existing evidence based protocols of care. | During acute care hospitalization

SECONDARY OUTCOMES:
Secondary outcome measures will be: length of stay, mortality, time to resolution and frequency of recurrence. | During acute care hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Etchells, MD MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada